CLINICAL TRIAL: NCT04728139
Title: Assessment of Glypican 3 as a Predictive Marker in Colorectal Cancer Patients
Brief Title: Assessment of Glypican 3 as Apredictive Marker in Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Hany Mohammed, residet doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: colorectal cancer
Record Dates: First submitted 2020-09-13; First posted 2021-01-28 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer
Keywords: glypican 3
MeSH Terms: conditions — Colorectal Neoplasms; Simpson-Golabi-Behmel syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with colorecta cancer (Active Comparator)
  Interventions: Diagnostic Test: glypican 3
- healthy individuals (No Intervention)

INTERVENTIONS:
Diagnostic Test: glypican 3 — Assessment of glypican 3 presence in colorectal cancer patients using ELISA
  Arms: patients with colorecta cancer

SUMMARY:
* Evaluation Of Glypican 3 in serum of colorectal cancer patients .
* Correlation between Glypican 3 and clinicopathological characteristics of colorectal cancer .

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy and the fourth most prominent cause of cancer-related deaths worldwide. Also it is the 7th commonest cancer in Egypt, representing 3.47% of male cancers and 3% of female cancers.The Glypicans , a family of proteins classified as HSPGs (heparan sulfate proteoglycan) , have been shown to interact with a number of growth factors and modulate growth factor activity and are linked to the xtracellular side of cell membrane by a glycosylphosphatidylinositol (GPI) anchor . Members of this large family of transmembrane proteins have been identified in both mammals and drosophila: 6 glypicans (GPC-1 through GPC-6) in mammals, and two others in the fly .Glypican-3 (GPC3) as one of this family is a protein of about 70 kD . It has multiple sugar chains and heparan sulfate modification sites . These proteins (Glypicans) participate in organ development by modulating extracellular growth signals and morphogen gradient formation, and are involved in human overgrowth and skeletal dysplasia problems .In some cancers, they are highly expressed, associated with tumorigenesis, and regulating angiogenesis for cancer progression and invasion . Abnormal expression of glypicans has been noted in multiple types of cancer. For examples, GPC-1 expression was found to be increased in breast cancer tissues and ovarian malignant tumors .GPC-2 is associated with neuroblastoma .Expression of GPC-3 was found in high-grade urothelial carcinoma and also reported in some non-CNS tumors of the brain.There have been several reports about the clinical usefulness of the N-terminal form of GPC3. Enzyme-linked immunosorbent assay methods capable of detecting the N-terminal form of GPC3 . A study of colorectal cancer tissue speciment shows a correlation between expression of GPC3 with the clinicopathologic variables such as the level of differentiation, GPC3 was found to be expressed in ( 42.8% ) of the well-differentiated tumors, and (50%) of the moderately differentiated tumors, (75%) of the moderately and poorly differentiated tumors .Therefore, it was found that the expression of GPC3 was correlated with the pathological grade of the tumors .

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer and admitted to south egypt cancer institute .

Exclusion Criteria:

* Other malignant diseases .
* Patients received chemotherapy for colorectal cancer .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Glypican 3 role as a predictive and diagnostic marker of colorectal marker . | 3 years
  measurment of GLYPICAN 3 level in serum of colorectal patients using ELISA method

SECONDARY OUTCOMES:
Addition of Glypican 3 to the routine markers of colorectal cancer . - Correlatin of this marker with the disease pathology and management procedures . | 3 years
  measurment of GLYPICAN 3 level in serum of colorectal patients using ELISA method

REFERENCES:
- [Background] Terzic J, Grivennikov S, Karin E, Karin M. Inflammation and colon cancer. Gastroenterology. 2010 Jun;138(6):2101-2114.e5. doi: 10.1053/j.gastro.2010.01.058. PMID 20420949
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Ijaz B, Formentin E, Ronci B, Locato V, Barizza E, Hyder MZ, Lo Schiavo F, Yasmin T. Salt tolerance in indica rice cell cultures depends on a fine tuning of ROS signalling and homeostasis. PLoS One. 2019 Apr 30;14(4):e0213986. doi: 10.1371/journal.pone.0213986. eCollection 2019. PMID 31039145
- [Background] Filmus J, Selleck SB. Glypicans: proteoglycans with a surprise. J Clin Invest. 2001 Aug;108(4):497-501. doi: 10.1172/JCI13712. No abstract available. PMID 11518720
- [Background] Shirakawa H, Kuronuma T, Nishimura Y, Hasebe T, Nakano M, Gotohda N, Takahashi S, Nakagohri T, Konishi M, Kobayashi N, Kinoshita T, Nakatsura T. Glypican-3 is a useful diagnostic marker for a component of hepatocellular carcinoma in human liver cancer. Int J Oncol. 2009 Mar;34(3):649-56. doi: 10.3892/ijo_00000190. PMID 19212669
- [Background] Sarrazin S, Lamanna WC, Esko JD. Heparan sulfate proteoglycans. Cold Spring Harb Perspect Biol. 2011 Jul 1;3(7):a004952. doi: 10.1101/cshperspect.a004952. PMID 21690215
- [Background] Fico A, Maina F, Dono R. Fine-tuning of cell signaling by glypicans. Cell Mol Life Sci. 2011 Mar;68(6):923-9. doi: 10.1007/s00018-007-7471-6. Epub 2011 Feb 22. PMID 18087675
- [Background] Matsuda K, Maruyama H, Guo F, Kleeff J, Itakura J, Matsumoto Y, Lander AD, Korc M. Glypican-1 is overexpressed in human breast cancer and modulates the mitogenic effects of multiple heparin-binding growth factors in breast cancer cells. Cancer Res. 2001 Jul 15;61(14):5562-9. PMID 11454708
- [Background] Davies EJ, Blackhall FH, Shanks JH, David G, McGown AT, Swindell R, Slade RJ, Martin-Hirsch P, Gallagher JT, Jayson GC. Distribution and clinical significance of heparan sulfate proteoglycans in ovarian cancer. Clin Cancer Res. 2004 Aug 1;10(15):5178-86. doi: 10.1158/1078-0432.CCR-03-0103. PMID 15297422
- [Background] Bosse KR, Raman P, Zhu Z, Lane M, Martinez D, Heitzeneder S, Rathi KS, Kendsersky NM, Randall M, Donovan L, Morrissy S, Sussman RT, Zhelev DV, Feng Y, Wang Y, Hwang J, Lopez G, Harenza JL, Wei JS, Pawel B, Bhatti T, Santi M, Ganguly A, Khan J, Marra MA, Taylor MD, Dimitrov DS, Mackall CL, Maris JM. Identification of GPC2 as an Oncoprotein and Candidate Immunotherapeutic Target in High-Risk Neuroblastoma. Cancer Cell. 2017 Sep 11;32(3):295-309.e12. doi: 10.1016/j.ccell.2017.08.003. PMID 28898695
- [Background] Aleksikova RIa. [On the morbidity of school-children in senior classes of Leningrad boarding schools]. Zdravookhr Ross Fed. 1965 Nov;9(11):11-3. No abstract available. Russian. PMID 4225756
- [Background] Chan ES, Pawel BR, Corao DA, Venneti S, Russo P, Santi M, Sullivan LM. Immunohistochemical expression of glypican-3 in pediatric tumors: an analysis of 414 cases. Pediatr Dev Pathol. 2013 Jul-Aug;16(4):272-7. doi: 10.2350/12-06-1216-OA.1. Epub 2013 Mar 26. PMID 23530909
- [Background] Haruyama Y, Yorita K, Yamaguchi T, Kitajima S, Amano J, Ohtomo T, Ohno A, Kondo K, Kataoka H. High preoperative levels of serum glypican-3 containing N-terminal subunit are associated with poor prognosis in patients with hepatocellular carcinoma after partial hepatectomy. Int J Cancer. 2015 Oct 1;137(7):1643-51. doi: 10.1002/ijc.29518. Epub 2015 Apr 6. PMID 25784484
- Available data/document: Study Protocol — http://rehamhany809@gmail.com